CLINICAL TRIAL: NCT04452357
Title: RT-155: Utilizing Pulsed Low-dose-rate (PLDR) Radiation to Prevent de Novo Stromal Activation; a Neoadjuvant Pancreatic Adenocarcinoma Phase I Trial
Brief Title: Pulse-low-dose Rate (PLDR) Radiation in Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-155; 18-1085 (Other: Fox Chase cancer Center)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PLDR Chemoradiation (Experimental): Patients will receive pulse-low-dose rate radiation, along with gemcitabine chemotherapy.
  6 patients each will be accrued at two dose levels. PLDR radiation will be delivered as 10 fractions of 20 cGy, initiated once every 3 minutes. Dose levels will be selected as follows: Dose level 1: 56 Gy; Dose level 2: 66 Gy
  Interventions: Radiation: PLDR

INTERVENTIONS:
Radiation: PLDR — PLDR radiation will be delivered as 10 fractions of 20 cGy, initiated once every 3 minutes. Dose levels will be selected as follows:
  Dose level 1: 56 Gy; Dose level 2: 66 Gy Drug: Gemcitabine

SUMMARY:
Standard chemoradiation, followed by surgery are standard treatment plan for patients suffering from pancreatic adenocarcinoma. Due to damage to the surrounding healthy tissue caused by standard radiation, this study uses a new type of radiation plan- pulsed low-dose rate (PLDR) radiation , in combination with chemotherapeutic drug, gemcitabine, given weekly along with the radiation.

DETAILED DESCRIPTION:
Radiation, combined with radiosensitizing chemotherapies, is often used preoperatively for borderline resectable cases with the intent of facilitating a curative surgical intervention. This includes providing margin adjacent to un-resectable vessels and sterilizing regional lymph nodes. Unfortunately, due to the radiosensitivity of adjacent small bowel and stomach, the total dose of radiation used is modest due to the risk of toxicities associated with higher doses. Pulsed low-dose-rate (PLDR) radiation improves the safety of radiation through breaking it up into small pulses. This increases the repair of DNA damage in normal tissues while remaining effective in cancer cells. Multiple prior studies have shown PLDR to be safe in the setting of re-irradiation, where additional radiation with conventional techniques is associated with severe toxicity.

PLDR radiation will be given in 2 doses to 6 patients at each dose level:

Dose level 1: 56 Gy- given over 6 weeks Dose level 2: 66 Gy- given over 7 weeks Standard chemotherapeutic drug, gemcitabine, will be administered once a week for the duration of radiation.

This treatment will be followed by standard surgery to remove the cancer after consultation with a surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically-confirmed pancreatic adenocarcinoma.
* Patients must have non-metastatic pancreatic cancer not appropriate for immediate surgical resection. This includes the following:

  * Any involvement (defined as loss of fat plane on contrast CT) of any of the following vessels*:

    * Common hepatic artery
    * Superior mesenteric artery
    * Celiac axis
    * Superior mesenteric vein
    * Portal vein
    * Aorta

      * These criteria will be judged by the operating surgeon in conjunction with a radiologist prior to enrollment.
  * Poor performance status not immediately conducive to radical surgery
  * Other clinical reasoning by the treating physicians that supports pre-operative chemoradiation
* Patients must have evaluable disease as measured by RECIST 1.1 criteria.
* Planned surgical resection at the time of enrollment (may be initially staged as resectable, borderline resectable, or locally-advanced/unresectable).
* Eastern Cooperative Oncology Group, or ECOG, performance status 0-2.
* Adequate bone marrow, hepatic, renal function.

  * ANC ³ 1,500/ml and PLT ³ 100,000/ml
  * Bilirubin less than 1.5 ULN
  * AST and ALT < 3X ULN
  * Serum Creatinine <1.5X ULN
* Prior chemotherapy allowed, but not mandatory. Patients who have undergone chemotherapy prior to participating in this study must have had a 2 week washout period at the time of signing the consent form.
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to registration. Postmenopausal woman must have been amenorrheic and nonlactating for at least 12 months to be considered of non-childbearing potential. Men and women of child bearing potential must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy is completed. Please refer to section 6.4 for additional detail.
* Age > 18 years
* Participants must sign a written informed consent and HIPAA consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.

Exclusion Criteria:

* Radiological or cytologically confirmed metastatic disease
* Patients who have had any prior therapy for pancreatic cancer, except chemotherapy (see 6.1.7)
* Concurrent non-study chemotherapy or biologic therapy
* A history of ataxia telangiectasia or other documented history of radiation hypersensitivity
* Scleroderma or active connective tissue disease
* Active inflammatory bowel disease
* Serious, active infections requiring treatment with IV antibiotics
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute grade 3+ gastrointestinal toxicity possibly, probably or definitely related to radiation. | 11 weeks
  Number of participants with Grade 3 toxicity related to the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States